CLINICAL TRIAL: NCT04609631
Title: Tai Chi for Comorbid Depression in T2DM Patients: A Randomized Controlled Trial Protocol
Brief Title: Tai Chi for Comorbid Depression in T2DM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Di Qin, Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019YFC1710302
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Depression; T2DM
Keywords: Tai Chi; Depression; T2DM; Randomized Controlled Trial
MeSH Terms: conditions — Depression | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tai Chi (5 times/week) (Experimental): 5 sessions of Tai Chi per week for 12 weeks
  Interventions: Behavioral: Tai Chi
- Tai Chi (3 times/week) (Experimental): 3 sessions of Tai Chi per week for 12 weeks
  Interventions: Behavioral: Tai Chi
- Tai Chi (1 time/week) (Experimental): 1 session of Tai Chi per week for 12 weeks
  Interventions: Behavioral: Tai Chi
- cognitive behavior therapy (CBT) (Active Comparator): 1 session of CBT per week for 12 weeks
  Interventions: Behavioral: CBT
- Waiting-list (No Intervention): Participants will maintain their routine treatment and life style for 12 weeks.

INTERVENTIONS:
Behavioral: Tai Chi — 24-form Tai Chi will be performed for 12 weeks. Each session contains a warm-up period (10 minutes), a Tai Chi period (40 minutes) and a cool-down period (10 minutes).
  Arms: Tai Chi (1 time/week); Tai Chi (3 times/week); Tai Chi (5 times/week)
Behavioral: CBT — CBT will be performed once a week for 12 weeks. Each session lasts for 1 hour.
  Arms: cognitive behavior therapy (CBT)

SUMMARY:
Previous studies suggested that Tai Chi may be beneficial for T2DM patients. However, no studies have investigated the effectiveness of Tai Chi for comorbid depression in T2DM patients, as well as the optimal frequency of Tai Chi. Thus, we intend to investigate the effectiveness of Tai Chi for comorbid depression in T2DM patients and test whether the effectiveness of Tai Chi depends on its frequency.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with depression by experienced psychiatrist;
* Participants diagnosed with T2DM by experienced endocrinologist;
* Participants aged between 18~75 years;
* Participants with HbA1c ranges from 6.5% to 8.5%;
* Participants with Hamilton Depression Scale (HAMD) (24-item-version) ranges from 20~35 scores;
* Participants passed the Physical Activity Readiness Questionnaire (PAR-Q);
* Participants willing to complete 12-week intervention and 12-week follow-up.
* Participants willing to sign informed consent form.

Exclusion Criteria:

* Participants with uncontrolled hypertension (SBP >160mmHg or DBP >100mmHg after taking hypotensive drugs);
* Participants with severe diabetic complications;
* Regular exercisers (at least 20 minutes/time, 3 times/week) in the last 3 months;
* Participants with cognitive impairment (Montreal Cognitive Assessment [MoCA] scores <26);
* Participants with history of bipolar disorder or schizophrenia or other mental illness;
* Participants with contraindications to exercise;
* Participants with acute, infectious diseases, cancer, or serious neurological disease, cardiovascular disease, pulmonary disease or other serious medical conditions limiting the ability;
* Participants taking psychoactive drugs;
* Participants participating in other clinical trials at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg depression rating scale | change from baseline to 12 weeks after intervention

SECONDARY OUTCOMES:
Montgomery Asberg depression rating scale | baseline, after intervention (12 weeks), after follow-up (24 weeks)
Hamilton Depression Scale (HAMD) (24-item-version) | change from baseline, after intervention (12 weeks), after follow-up (24 weeks)
Social Disability Screening Schedule | baseline, after intervention (12 weeks), after follow-up (24 weeks)
EuroQol-5D questionnaire | baseline, after intervention (12 weeks), after follow-up (24 weeks)
Clinical Global Impression scale | after intervention (12 weeks), after follow-up (24 weeks)
Biochemical indicators | baseline, after intervention (12 weeks), after follow-up (24 weeks)
  HbA1c
Fasting plasma glucose | baseline, after intervention (12 weeks), after follow-up (24 weeks)
  Biochemical indicators
Postprandial plasma glucose | baseline, after intervention (12 weeks), after follow-up (24 weeks)
  Biochemical indicators
insulin level | baseline, after intervention (12 weeks), after follow-up (24 weeks)
  Biochemical indicators

OTHER OUTCOMES:
Pittsburgh sleep quality index | baseline, after intervention (12 weeks), after follow-up (24 weeks)
Hamilton Anxiety Rating Scale | baseline, after intervention (12 weeks), after follow-up (24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Youping Liu, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Henan University of Chinese Medicine, Zhengzhou, Henan
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine (Sichuan Provincial Hospital of Traditional Chinese Medicine), Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No